CLINICAL TRIAL: NCT02340364
Title: Patient NAVIgation to Reduce Readmissions Among Black Men With Heart Disease
Acronym: NAVI-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Reagan W. Durant, MD, Principal investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: X130515002
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Heart Diseases
Keywords: Hospital Readmissions; Patient Navigation
MeSH Terms: conditions — Heart Diseases | interventions — Educational Status; Patient Navigation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education + PN Arm (Experimental): 208 patients randomized to self-care education+ Patient navigator-delivered self-care plan.
  Interventions: Behavioral: Education + Patient Navigation
- Educational Control Arm (Active Comparator): - 208 patients randomized to self-care education alone.
  Interventions: Behavioral: Self-care Education

INTERVENTIONS:
Behavioral: Education + Patient Navigation — 208 patients randomized to self-care Education+ Patient Navigation-delivered self-care plan.
  Arms: Education + PN Arm
Behavioral: Self-care Education — 208 patients randomized to self-care education alone.
  Arms: Educational Control Arm

SUMMARY:
The investigators are asking subjects to take part in the Patient NAVIgation to Reduce Readmissions among Black Men with Heart Disease (NAVI-HF) research study. This research study will test how well trained laypeople working as patient navigators will help patients recently hospitalized for heart failure avoid future hospitalizations. NAVI-HF is a new program sponsored by funding from the National Institute of Minority Health and Health Disparities. People who enter into the study will work with a patient navigator to undergo the full program or work with a trained layperson to receive general education on heart disease treatment and prevention. The purpose of the study is to determine whether a patient navigation program will be effective in reducing the number of hospitalizations in the future for program participants. This study will enroll 416 participants from UAB.

DETAILED DESCRIPTION:
Therefore, in the Patient NAVIgation to Reduce Readmissions among Black Men with Heart Disease (NAVI-HF) study, the investigators propose to recruit 416 AA men with Heart Disease receiving inpatient care at UAB Hospital and randomize them either to Heart Disease self-care education plus a patient navigator-delivered self-care plan (Education + PN arm) or to Heart Disease self-care education alone (Educational Control arm). The investigators will compare participant outcomes such as all-cause and Heart Disease readmission rates, Heart Disease self-care adherence as well as cost effectiveness across the two intervention arms. Our Specific Aims are:

1. To assess the 30-day all-cause readmission rates among male African American Heart Disease patients receiving Heart Disease self-care education plus a patient navigator-delivered self-care plan versus Heart Disease self-care education alone
2. To assess the Heart Disease self-efficacy and heart failure self-care adherence among male African American Heart Disease patients receiving Heart Disease self-care education plus a patient navigator-delivered self-care plan versus Heart Disease self-care education alone
3. To evaluate the cost-effectiveness of Heart Disease self-care education plus a patient navigator-delivered self-care plan versus Heart Disease self-care education alone

ELIGIBILITY:
Inclusion Criteria:

* African American
* Male
* Age = 30 or older
* Inpatient admission at UAB Hospital or UAB Medical West with a diagnosis of heart disease as a principle or one of the first 3 diagnosis.
* Residence in Jefferson or Shelby Counties, Alabama within 45 miles of UAB Hospital.
* English Speaking
* Physically and cognitively able to listen to 30-minute video undergo a home visit and telephone contacts over several weeks.

Exclusion Criteria:

* Heart transplant or awaiting heart transplant (admitted to UAB Advanced HF/Transplant Service).
* Currently participating in another clinical research study with an overlapping intervention.
* Current or anticipated long term (>2 weeks) residence in a skilled nursing facility.
* Patients who indicated that they were unwilling to make lifestyle changes now or in the near future.
* Patients whose symptoms may be eliminated by surgery (e.g., severe aortic stenosis) or who had undergone surgery (e.g., coronary artery bypass grafting valvular replacement/repair) in the last month.

Ages: 30 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2015-03; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Readmission Rates | Within 30 days
  Re-hospitalization of Heart Disease patients within 30 days of being discharged home.

CONTACTS AND LOCATIONS:
Overall Officials: Raegan W Durant, M.D., MPH, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - UAB Medical West, Bessemer, Alabama
  - UAB, Birmingham, Alabama